CLINICAL TRIAL: NCT05142124
Title: German Cardiac Arrest Registry
Acronym: G-CAR
Status: Recruiting | Type: Observational
Sponsor: Leipzig Heart Science gGmbH (Other)
Collaborators: Helios Health Institute GmbH (Other); Heart Center Leipzig - University Hospital (Other); IHF GmbH - Institut für Herzinfarktforschung (Other); Universitätsklinikum Hamburg-Eppendorf (Other); St. Antonius Hospital (Other); Klinikum Ludwigshafen (Other); University of Magdeburg (Other); Charite University, Berlin, Germany (Other); University Hospital of Cologne (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-0396
Record Dates: First submitted 2021-11-08; First posted 2021-12-02 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Out-of-hospital Cardiac Arrest
Keywords: Out-of-hospital Cardiac Arrest; OHCA; resuscitation; cardiac arrest center; acute care medicine; intensive care; post-resuscitation care
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In Germany, 70.000 to 100.000 patients suffer from out-of-hospital cardiac arrest (OHCA) every year. More than half of these are due to cardiac causes. Despite the medical progress over the last decades, rates of survival with good neurological outcome remain low. For many below-mentioned issues, no adequate evidence from randomized trials is available. Therefore, a systematic and standardized recording of the pre-clinical, clinical and post-clinical treatment course and of the clinical outcomes of OHCA patients is essential to improve patient care. Aim of the German Cardiac Arrest Registry (G-CAR) is to achieve a better understanding of the disease entity, leading to an optimized treatment of OHCA patients. The recorded data include information on demographic and psychosocial aspects, course of the disease, clinical, laboratory and other examinations as well as treatment modalities in patients with OHCA due to a cardiac cause.

ELIGIBILITY:
Inclusion Criteria:

* patients with out-of-hospital cardiac arrest with assumed cardiovascular cause

Exclusion Criteria:

* rejection of register participation by patient or legal representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with out-of-hospital cardiac arrest with assumed cardiovacular cause
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
In hospital mortality | until discharge, an average of 2 weeks

SECONDARY OUTCOMES:
Length of ICU stay | until discharge, an average of 2 weeks
Length of hospital stay | until discharge, an average of 2 weeks
Mortality | Day 30
Mortality | Month 6
European Quality of Life 5 Dimensions 5 Level Version (EQ-5D) | Month 6
  five levels in each dimension are worded as (1) 'not /no problems', (2) 'slight problems', (3) 'moderate problems', (4) 'severe problems', and (5) 'unable to'
Post Traumatic Stress Syndrome | Month 6
  PTSS-14
Reintegration | Month 6
  Reintegration to Normal Living Index
Hospital Anxiety and Depression Scale (HADS) | Month 6
  score 0-21; higher value show more severe depression
Mini Montreal Cognitive Assessment (MoCA) | Month 6
  score 0-15; 11 or higher is normal, 10 or less indicate cognitive dysfunction
Mini Montreal Cognitive Assessment (MoCA) | Month 12
  score 0-15; 11 or higher is normal, 10 or less indicate cognitive dysfunction
Mortality | Month 12
European Quality of Life 5 Dimensions 5 Level Version (EQ-5D) | Month 12
  five levels in each dimension are worded as (1) 'not /no problems', (2) 'slight problems', (3) 'moderate problems', (4) 'severe problems', and (5) 'unable to'
Post Traumatic Stress Syndrome (PTSS-14) | Month 12
  scor 14-98; higher value indicate more post traumatic stress
Reintegration | Month 12
  Reintegration to Normal Living Index
Hospital Anxiety and Depression Scale (HADS) | Month 12
  score 0-21; higher value indicate more severe depression

CONTACTS AND LOCATIONS:
Overall Officials: Janine Pöss, Dr., Study Chair — Heart Center Leipzig at University of Leipzig, Department of Internal Medicine/Cardiology
Locations (25):
- Germany (25):
  - CHARITE - Universitätsmedizin Berlin - Campus Virchow Klinikum, Berlin, State of Berlin
  - SLK-Kliniken Heilbronn - Klinikum am Plattenwald, Bad Friedrichshall
  - Charité Universitätsmedizin Berlin - Deutsches Herzzentrum Berlin, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Bremer Institut für Herz- und Kreislaufforschung am Klinikum Links der Weser, Bremen
  - Herzzentrum der Universität zu Köln, Cologne
  - Herzzentrum Dresden GmbH, Dresden
  - Universitätsklinikum Düsseldorf - Klinik für Kardiologie, Pneumologie und Angiologie, Düsseldorf
  - Elisabeth Krankenhaus Essen - Klinik für Akut- und Notfallmedizin, Essen
  - Klinikum Frankfurt Höchst, Frankfurt
  - Universitätsklinikum Halle (Saale), Halle
  - Universitäres Herz- und Gefäßzentrum Hamburg, Hamburg
  - Asklepios Klinik St- Georg Hamburg, Hamburg
  - SLK-Kliniken Heilbronn - Klinikum am Gesundbrunnen, Heilbronn
  - Universitätsklinikum des Saarlandes, Homburg
  - Heart Center Leipzig at University of Leipzig, Department of Internal Medicine/Cardiology, Leipzig
  - Klinikum der Stadt Ludwigshafen gGmbH, Ludwigshafen
  - Herzzentrum Lübeck, Lübeck
  - Universitätsklinikum Mannheim, Mannheim
  - Klinikum der Universität München, München
  - Marienhaus Klinikum Hetzelstift, Neustadt
  - Hegau-Bodensee Klinikum, Singen
  - Hegau-Bodensee-Klinikum Singen, Singen
  - Schwarzwald-Baar Klinikum VS, Villingen-Schwenningen
  - Dr. Horst Schmidt Kliniken, Wiesbaden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Poss J, Sinning C, Rossberg M, Hosler N, Ouarrak T, Bottiger BW, Ewen S, Wienbergen H, Voss F, Dutzmann J, Tigges E, Voigt I, Freund A, Desch S, Michels G, Thiele H, Zeymer U; G-CAR Investigators. German Cardiac Arrest Registry (G-CAR)-results of the pilot phase. Clin Res Cardiol. 2025 Oct;114(10):1270-1279. doi: 10.1007/s00392-024-02468-5. Epub 2024 Jun 13. PMID 38869632
- [Derived] Poss J, Sinning C, Schreiner I, Apfelbacher C, Drewitz KP, Hosler N, Schneider S, Pieske B, Bottiger BW, Ewen S, Wienbergen H, Kelm M, Bock D, Graf T, Adler C, Dutzmann J, Knie W, Orban M, Zeymer U, Michels G, Thiele H; G-CAR Investigators. German Cardiac Arrest Registry: rationale and design of G-CAR. Clin Res Cardiol. 2023 Apr;112(4):455-463. doi: 10.1007/s00392-022-02044-9. Epub 2022 Jun 21. PMID 35729429